CLINICAL TRIAL: NCT04004390
Title: Treatment of Post-poliomyelitis Syndrome by Intravenous Immunoglobulin: a Retrospective Study of Efficacy on Clinical and Isokinetic Criteria
Brief Title: Treatment of Post-poliomyelitis Syndrome by Intravenous Immunoglobulin
Acronym: PPS and IGIV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0322
Record Dates: First submitted 2019-06-28; First posted 2019-07-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Post-Poliomyélitis Syndrom
Keywords: Pre- and post-therapeutic evaluation carried out; Data transcribed in the computerized patient file; post-poliomyelitis syndrome; Intravenous immunoglobulins; walking test; isokinetics
MeSH Terms: conditions — Postpoliomyelitis Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our study evaluates the efficacy of IGIV treatment in PPS on clinical (walking and pain) and isokinetic (muscle strength) criteria, on patients with PS at Montpellier's Hospital

DETAILED DESCRIPTION:
Patients are admitted to a multidisciplinary consultation (neurologist, PMK) to validate the indication of treatment with IGIV. Realization of a pre-therapeutic evaluation in the department of MPR on the criteria of judgment, then the patient is admitted in a service of neurology to benefit from the cure of IGIV. The patient is then re-admitted to a PMR service for post-treatment evaluation.

Collection of data retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPS
* Pre- and post-therapeutic evaluation carried out
* Data transcribed in the computerized patient file

Exclusion Criteria:

* No walking patient

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 men and 11 women with Diagnosis of PPS
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Muscular strength | 5 months
  Muscular strength with isokinetic

SECONDARY OUTCOMES:
Walking perimeter | 5 months
  Walking perimeter with walking test (6 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: MOIZIARD Vincent, intern, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC